CLINICAL TRIAL: NCT00882596
Title: A Multi-Site, Prospective, Non-Randomized Study of the Contura™ Multi-Lumen Balloon (MLB) Catheter to Deliver Accelerated Partial Breast Irradiation: Analysis of Dosimetry, Local Tumor Control, Cosmetic Outcome, and Toxicity
Brief Title: Use of the Contura™ Catheter to Deliver Accelerated Partial Breast Irradiation to "Low-risk" Breast Cancer Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cancer Center of Irvine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S07-002; 1098558
Record Dates: First submitted 2009-04-15; First posted 2009-04-16 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Breast Cancer
Keywords: Contura; Cancer; Accelerated; Partial; Breast; Irradiation
MeSH Terms: conditions — Breast Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Contura accelerated partial breast irradiation. Following a lumpectomy, a Contura balloon catheter is placed in the lumpectomy cavity. Later that morning, accelerated partial breast irradiation begins.
  Interventions: Device: Accelerated partial breast irradiation

INTERVENTIONS:
Device: Accelerated partial breast irradiation — A total radiation dose of 34 Gy is delivered in 10 fractions bid over 5-7 days with 6 hours between the radiation treatments each day. Each radiation treatment takes 15-30 minutes. There is no radioactivity left behind in the patient.
  Other Names: Contura catheter

SUMMARY:
The purpose of this national, multi-site study is to determine the safety and effectiveness of the Contura catheter in breast cancer patients undergoing accelerated partial breast irradiation.

DETAILED DESCRIPTION:
The Cancer Center of Irvine is one of the busiest centers in the United States for Contura accelerated partial breast irradiation.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to sign informed consent
* Age 50 or older at diagnosis
* Life expectancy greater than 10 years (excluding diagnosis of breast cancer)
* Surgical treatment of the breast must have been lumpectomy. The margins of the resected specimen must be histologically free of tumor (negative surgical margins per NSABP criteria)
* On histologic examination, the tumor must be DCIS and/or invasive breast carcinoma
* For patients with invasive breast cancer, an axillary staging procedure must be performed [either sentinel node biopsy or axillary dissection (with a minimum of 6 axillary nodes removed), and the axillary node(s) must be pathologically negative]
* The T stage must be Tis, T1, or T2. If T2, the tumor must be less than or equal to 3.0 cm in maximum diameter
* Estrogen receptor positive tumor

Exclusion Criteria:

* Age < 50 at diagnosis (regardless of histology)
* Pregnant or breast-feeding
* Active collagen vascular disease
* Paget's disease of the breast
* Prior history of DCIS or invasive breast cancer
* Prior breast or thoracic radiation therapy for any condition
* Multicentric carcinoma (DCIS or invasive)
* Synchronous bilateral invasive or non-invasive breast cancer
* Surgical margins that cannot be microscopically assessed or that are positive
* Positive axillary node(s)
* T stage of T2 with the tumor > 3 cm in maximum diameter or a T stage of T3 or T4
* Estrogen receptor negative tumor

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-05; Primary Completion 2013-05 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Maximum total skin dose is less than or equal to 125% of the prescribed radiation dose. | 19 months

SECONDARY OUTCOMES:
Toxicity rates | 79 months

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth M Tokita, MD, Principal Investigator — Cancer Center of Irvine; Richard B Wilder, MD, Study Director — Cancer Center of Irvine
Locations (1):
- Cancer Center of Irvine, Irvine, California, United States